CLINICAL TRIAL: NCT03454451
Title: A PHASE 1/1b MULTICENTER STUDY TO EVALUATE THE HUMANIZED ANTI-CD73 ANTIBODY, CPI-006, AS A SINGLE AGENT OR IN COMBINATION WITH CIFORADENANT, WITH PEMBROLIZUMAB, AND WITH CIFORADENANT PLUS PEMBROLIZUMAB IN ADULT SUBJECTS WITH ADVANCED CANCERS
Brief Title: CPI-006 Alone and in Combination With Ciforadenant and With Pembrolizumab for Patients With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corvus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPI-006-001
Record Dates: First submitted 2018-02-05; First posted 2018-03-06 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Non-Small Cell Lung Cancer; Renal Cell Cancer; Colorectal Cancer; Triple Negative Breast Cancer; Cervical Cancer; Ovarian Cancer; Pancreatic Cancer; Endometrial Cancer; Sarcoma; Squamous Cell Carcinoma of the Head and Neck; Bladder Cancer; Metastatic Castration Resistant Prostate Cancer; Non-hodgkin Lymphoma
Keywords: NSCLC; RCC; TNBC; mCRPC; CRC; Lung Cancer; Kidney Cancer; Rectal Cancer; Breast Cancer; Sarcoma; Endometrial; Pancreatic; Ovarian; SCCHN; NHL
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Colorectal Neoplasms; Triple Negative Breast Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Endometrial Neoplasms; Sarcoma; Squamous Cell Carcinoma of Head and Neck; Urinary Bladder Neoplasms; Lymphoma, Non-Hodgkin; Lung Neoplasms; Kidney Neoplasms; Rectal Neoplasms; Breast Neoplasms | interventions — CPI-006; ciforadenant; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1a (Experimental): CPI-006
  Interventions: Drug: CPI-006
- Cohort1b (Experimental): CPI-006 + ciforadenant
  Interventions: Drug: CPI-006 + ciforadenant
- Cohort 1c (Experimental): CPI-006 + pembrolizumab
  Interventions: Drug: CPI-006 + pembrolizumab
- Cohort 2a (Experimental): CPI-006
  Interventions: Drug: CPI-006
- Cohort 2b (Experimental): CPI-006 + ciforadenant
  Interventions: Drug: CPI-006 + ciforadenant
- Cohort 2c (Experimental): CPI-006 + pembrolizumab
  Interventions: Drug: CPI-006 + pembrolizumab

INTERVENTIONS:
Drug: CPI-006 — Subjects will receive escalating doses of CPI-006 administered intravenously once every 21 days until MTD is reached or until disease progression.
  Arms: Cohort 1a
Drug: CPI-006 + ciforadenant — Subjects will receive escalating doses of CPI-006 administered intravenously once every 21 days in combination with CPI-444 orally twice daily until MTD is reached for CPI-006 or until disease progression.
  Arms: Cohort1b
Drug: CPI-006 + pembrolizumab — Subjects will receive escalating doses of CPI-006 in combination with pembrolizumab administered intravenously once every 21 days until MTD is reached for CPI-006 or until disease progression.
  Arms: Cohort 1c
Drug: CPI-006 — Selected dose of CPI-006 administered intravenously once every 21 days until disease progression.
  Arms: Cohort 2a
Drug: CPI-006 + ciforadenant — Selected dose of CPI-006 administered intravenously once every 21 days, in combination with CPI-444 orally twice daily until disease progression.
  Arms: Cohort 2b
Drug: CPI-006 + pembrolizumab — Selected dose of CPI-006 in combination with pembrolizumab administered intravenously once every 21 days until disease progression.
  Arms: Cohort 2c

SUMMARY:
This is a Phase 1/1b open-label, dose escalation and dose expansion study of CPI-006, a humanized monoclonal antibody (mAb) targeting the CD73 cell-surface ectonucleotidase in adult subjects with select advanced cancers. CPI-006 will be evaluated as a single agent, in combination with ciforadenant (an oral adenosine 2A receptor antagonist), in combination with pembrolizumab (an anti-PD1 antibody), and in combination with ciforadenant and pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
2. Documented incurable cancer with one of the following histologies: nonsmall cell lung cancer, renal cell cancer, triple negative breast cancer, colorectal cancer with microsatellite instability(MSI), bladder cancer, cervical cancer, uterine cancer, sarcoma, endometrial cancer, and metastatic castration resistant prostate cancer.
3. At least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
4. For Escalation: At least 1 but not more than 5 prior systemic therapies for advanced/ recurrent or progressing disease. For Expansion: Subject must have progressed on, be refractory to, or intolerant to 1-3 prior systemic therapies.
5. Willingness to provide tumor biopsies.

Exclusion Criteria

1. History of severe hypersensitivity reaction to monoclonal antibodies.
2. Subjects who have received prior therapy with regimens containing cytotoxicT-lymphocyte antigen-4 (CTLA-4), programmed cell death ligand 1 (PDL1), or PD1 antagonists are NOT permitted to enroll unless all adverse events (AEs) while receiving prior immunotherapy have resolved to Grade 1 or baseline prior to screening.
3. History of (non-infectious) pneumonitis that required steroids or subject has current pneumonitis.
4. The use of any investigational medication or device in the 30 days prior to screening and throughout the study is prohibited.
5. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-02-19 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) of CPI-006 as a single agent and in combination with ciforadenant and with pembrolizumab. | From start of treatment to end of treatment, up to 36 months
Incidence of treatment-emergent adverse events as assessed by NCI CTCAE v.4.03, of CPI-006 as single agent and in combination with ciforadenant and with pembrolizumab. | From start of treatment to end of treatment, up to 36 months
Identify the MDL(maximum dose level) of single agent CPI-006 | From start of treatment to end of treatment, up to 36 months

SECONDARY OUTCOMES:
Area under the curve (AUC) of CPI-006 | Day 1, 2, 8 , and 15 of Cycle 1 & 4 (each cycle is 21 days).
Maximum serum concentration (Cmax) of CPI-006 | Day 1, 2, 8 , and 15 of Cycle 1 & 4 (each cycle is 21 days).
Objective response rate per RECIST v.1.1 criteria of CPI-006 as single agent and in combination with ciforadenant and with pembrolizumab. | From start of treatment to end of treatment, up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: S Mahabhashyam, MD, Study Chair — Corvus Pharmaceuticals
Locations (27):
- United States (22):
  - Arizona Oncology, Tucson, Arizona
  - City Of Hope, Duarte, California
  - UC San Francisco, San Francisco, California
  - Yale School of Medicine, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - The John Hopkins University, Baltimore, Maryland
  - Dana Farber, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - NY Hematology, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Carolina BioOncology Institute, Huntsville, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - University of Oklahoma - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - UPMC Hillman, Pittsburgh, Pennsylvania
  - Greenville, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - Virginia Cancer, Fairfax, Virginia
  - Froedtert Hospital & Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Lifehouse, Camperdown, New South Wales
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Westmead, Westmead, New South Wales
  - Royal Brisbane, Herston, Queensland
  - Monash Hospital, Clayton, Victoria

REFERENCES:
- [Derived] Miller RA, Luke JJ, Hu S, Mahabhashyam S, Jones WB, Marron T, Merchan JR, Hughes BGM, Willingham SB. Anti-CD73 antibody activates human B cells, enhances humoral responses and induces redistribution of B cells in patients with cancer. J Immunother Cancer. 2022 Dec;10(12):e005802. doi: 10.1136/jitc-2022-005802. PMID 36600561